CLINICAL TRIAL: NCT00002224
Title: Comparison of HIV RNA Suppression Produced by Triple Regimens Containing Either Didanosine Enteric Coated or Didanosine Formulations Each Administered Once Daily
Brief Title: Comparison of Two Anti-HIV Regimens That Include One of Two Forms of Didanosine (ddI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 039G; AI454-158
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Drug Administration Schedule; Stavudine; HIV Protease Inhibitors; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
Didanosine is an effective anti-HIV drug, but it can cause stomach upset. This study tests a new form of didanosine, ddI EC, a coated pill that passes through the stomach more easily and hopefully will prevent stomach upset. The purpose of this study is to compare the effectiveness of ddI EC versus the standard form of ddI. Both forms of ddI will be given with stavudine (d4T) plus nelfinavir (NLF).

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 open-label treatment groups. Group 1 receives ddI EC plus d4T plus NLF for 48 weeks. Group 2 receives ddI plus d4T plus NLF for 48 weeks. Both forms of ddI are administered orally once daily. Antiviral activity is determined by the magnitude and the duration of reduction of plasma HIV RNA from baseline through Week 24.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 18 years old.
* Have a viral load of at least 5,000 copies/ml and a CD4 count of at least 100 cells/mm3.

Exclusion Criteria

You will not be eligible for this study if you:

* Have received more than 4 weeks of treatment with nucleoside anti-HIV medications (NRTIs), or more than 1 week with protease inhibitors. (All anti-HIV treatments other than study medications must be stopped at least 14 days prior to study entry.)
* Have severe diarrhea.
* Are pregnant or breast-feeding.
* Have a history of pancreatic disease or any other serious condition.
* Have hepatitis within 30 days prior to study entry.
* Cannot take medications by mouth.
* Have received certain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1999-03; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (22):
  - Sorra Research Ctr / Med Forum, Birmingham, Alabama
  - AIDS Healthcare Foundation, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - Beacon Clinic / Boulder Community Hosp, Boulder, Colorado
  - Community Health Care, Fort Lauderdale, Florida
  - Immunity Care and Research Inc, Fort Lauderdale, Florida
  - HIV Clinical Research Ctr, Fort Lauderdale, Florida
  - South Shore Hosp, Miami, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Clinical Studies of Las Vegas, Las Vegas, Nevada
  - Anderson Clinical Research Inc, Rego Park, New York
  - Anderson Clinical Research Inc, Reading, Pennsylvania
  - Coastal Carolina Research Ctr, Mt. Pleasant, South Carolina
  - Oak Lawn Physicians Group, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Nicholaos Bellos, Dallas, Texas
  - Houston Clinical Research Network / Div of Montrose Clinic, Houston, Texas
  - Swedish Med Ctr, Seattle, Washington
- Canada (2):
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec